CLINICAL TRIAL: NCT02343952
Title: A Phase II Trial of Concurrent Chemoradiation With Consolidation Pembrolizumab for the Treatment of Inoperable or Unresectable Stage III Non-Small Cell Lung Cancer (NSCLC): HCRN LUN14-179
Brief Title: Consolidation Pembrolizumab Following Chemoradiation in Patients With Inoperable/Unresectable Stage III NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN14-179
Record Dates: First submitted 2015-01-06; First posted 2015-01-22 (Estimated); Results first posted 2022-01-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Pembrolizumab; MK-3475
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental): Pembrolizumab -200 mg IV 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab, 200 mg IV every 3 weeks (until PD, unacceptable toxicity, or after 12 months of therapy with pembrolizumab.
  Other Names: MK-3475

SUMMARY:
This is an open label, multi-institutional, single arm phase II trial of consolidation therapy with pembrolizumab, following initial treatment with concurrent chemoradiation in patients with inoperable or unresectable stage IIIA or IIIB NSCLC. No randomization or blinding is involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Eligible patients must have completed concurrent chemoradiation with a standard chemotherapy regimen (either cisplatin/etoposide or carboplatin/paclitaxel) and a dose of radiation ranging from 59.4-66.6Gy, with restaging completed 28 days to 56 days post-chemoradiation. Patients with progressive disease will not be eligible for investigational treatment. Patients with stable disease/response will be eligible to register for investigational treatment of consolidation therapy to begin a minimum of 28 days and a maximum of 56 days from completion of chemoradiotherapy.

INVESTIGATIONAL TREATMENT:

Pembrolizumab, 200 mg IV every 3 weeks (until progressive disease (PD), unacceptable toxicity, or after 12 months (52 weeks) of therapy with pembrolizumab.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Hematopoietic:

* Absolute neutrophil count (ANC) ≥1,500/mcL
* Platelets ≥100,000/mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L

Renal:

* Serum creatinine OR measured or calculated creatinine clearance ≤1.5 X institutional upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl)

Hepatic:

* Serum total bilirubin ≤ 1.5 X institutional ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 institutional ULN
* Aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT), alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 X institutional ULN

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X institutional ULN unless subject is receiving anticoagulant therapy as long as PT/INR/PTT is within therapeutic range of intended use of anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of NSCLC
* Must have unresectable or inoperable stage IIIA or IIIB disease. Patients are considered unresectable or inoperable based on the judgment of the treating physician
* Must have completed concurrent chemoradiation with a standard chemotherapy regimen (either cisplatin/etoposide or carboplatin/paclitaxel) and a dose of radiation ranging from 59.4-66.6Gy
* Must have stable disease or disease response as evidenced on CT evaluation a minimum of 28 days and a maximum of 56 days following the completion of chemoradiation
* Women of childbearing potential must be willing to use two methods of contraception or abstain from heterosexual activity from the point of registration through 120 days after the last dose of study drug
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of the study drug through 120 days after the last dose of the study drug
* Age ≥ 18 years at the time of consent
* Written informed consent and HIPAA authorization for release of personal health information

Exclusion Criteria:

* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Active central nervous system (CNS) metastases. Subjects must undergo a head computed tomography (CT) scan or brain MRI within 28 days prior to registration for protocol therapy to exclude brain metastases if symptomatic or without prior brain imaging
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy
* Prior chemotherapy, adjuvant therapy, or radiotherapy for lung cancer, other than standard concurrent chemoradiation as described above
* Prior therapy with a PD-1, PD-L1, or CTLA-4 inhibitor or a lung cancer-specific vaccine therapy
* Presence of metastatic disease (stage IV NSCLC) is not allowed. Subjects must be evaluated with a PET scan within 28 days prior to registration for protocol therapy to exclude metastatic disease
* No active second cancers
* Evidence of active autoimmune disease requiring systemic treatment within the past 90 days or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids
* Diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy or other immunosuppressive therapy (excludes inhaled corticosteroids) within 7 days of first dose of study drug
* History of psychiatric illness or social situations that would limit compliance with study requirements
* Clinically active infection as judged by the treating investigator (≥ Grade 2 by CTCAE v4) including known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Cancer Research Network
Locations (15):
- United States (15):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Fort Wayne Oncology & Hematology, Inc., Fort Wayne, Indiana
  - IU Health Goshen Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - IU Health at Ball Memorial Hospital, Muncie, Indiana
  - Oncology Hematology Associates of SW Indiana, Newburgh, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Study Treatment
Arm/Group | Experimental Arm
Started | 93
Completed | 40
Not Completed | 53
Not completed — Disease Progression | 23
Not completed — Death | 3
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 7
Not completed — other complicating Diseases | 1
Period: Follow up
Arm/Group | Experimental Arm
Started | 83
Completed | 38
Not Completed | 45
Not completed — Withdrawal by Subject | 3
Not completed — Death | 33
Not completed — Patient does not meet eligibility for study. | 1
Not completed — Research department closed by the practice. | 5
Not completed — Patient went home to Russia | 1
Not completed — Disease Progression | 1
Not completed — study terminated | 1

BASELINE CHARACTERISTICS:
Population: This includes all subjects with exception of one subject.This patient had change in diagnosis from non-small cell carcinoma to uterine adenocarcinoma while on study. In retrospect, patient does not meet eligibility for study. Therefore, this subject was included in the safety results, but not the efficacy results.
Arm/Group | Experimental Arm
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 84
  Race: Black or African American | 3
  Race: Asian | 4
  Race: Unknown | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic | 90
  Ethnicity: Unknown | 2
Disease Stage [Count of Participants; unit: Participants] — Stage IIIA includes smaller tumors (T1-T2) associated with ipsilateral bronchopulmonary, and hilar (N1) or mediastinal (N2) lymph node involvement, as well as large, locally invasive tumors (T3 or T4) when associated with N0 or N1. At the next level, stage IIIB includes tumors associated with spread to contralateral mediastinal or supraclavicular lymph nodes (N3), exactly like T3 or T4 tumors with N2.
  The average overall survival time in subjects at stage IIIA NSCLC is 22.930 months whereas at stage IIIB is 23.081 months.
  Participants
    IIIA | 55
    IIIB | 37
Tumor Histologic Type [Count of Participants; unit: Participants]
  Squamous | 41
  Non-Squamous | 51
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 16
  Former smoker | 71
  Never smoker | 5
Prior Radiation Dose [Mean (Standard Deviation); unit: Gray] | 61.0 (6.2)
Prior Chemo Received [Count of Participants; unit: Participants]
  Cisplatin/Etoposide | 24
  Carboplatin/Paclitaxel | 65
  Cisplatin/Pemetrexed | 2
  Carboplatin/Paclitaxel & Carboplatin/Pemetrexed | 1
PD-L1 [Count of Participants; unit: Participants]
  Negative | 11
  Positive(1-49%) | 11
  Positive(>=50%) | 31
  Missing/Not collected | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Death or Distant Metastasis
Description: Time to Death or Distant Metastasis is defined as the time from the date of randomization until the first date of distant metastasis or death in the absence of distant metastasis. Distant metastasis is defined as any new lesion that was outside of the radiation field according to RECIST 1.1 or proven by biopsy. The Primary objective in the study was to determine if consolidation therapy with pembrolizumab following concurrent chemoradiation improves time to death or distant metastatic disease, depending on which occurs first, in subjects with inoperable or unresectable stage IIIA or IIIB NSCLC.
Time Frame: From start of treatment until death or distant metastasis (estimate 18 months) up to a maximum of 47 months.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 92
months | 30.7 [18.7 to NA] — The upper limit of the confidence interval was not reached.

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from randomization until the date of objective disease progression (RECIST 1.1) or death (by any cause in the absence of progression). Progression is defined using RECIST 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. One of the secondary objectives in the study is to determine if consolidation therapy with pembrolizumab following concurrent chemoradiation improves progression free survival in subjects with inoperable or unresectable stage IIA or IIIB non-small cell lung cancer(NSCLC). PFS has been estimated by Kaplan-Meier method.
Time Frame: From start of treatment until Progression based on RECIST 1.1 or death up to a maximum value of 47 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 92
months | 18.7 [12.4 to 33.8]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the date of randomization until death due to any cause. One of the secondary objectives in the study is to determine if consolidation therapy with pembrolizumab following concurrent chemoradiation improves Overall Survival in subjects with inoperable or unresectable stage IIA or IIIB non-small cell lung cancer(NSCLC). OS has been estimated by Kaplan-Meier method.
Time Frame: From the date of randomization up to a maximum value of 47 months or death.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm
Number analyzed (Participants) | 92
months | 35.8 [24.2 to NA] — The upper limit of the confidence interval was not reached.

4. Secondary Outcome: Number of Participants Experiencing Grade 3-4 AE With Adverse Events as a Measure of Safety and Tolerability
Description: One of the secondary objective in this study is to assess toxicity and tolerability of pembrolizumab consolidation therapy following concurrent chemoradiation in subjects with stage IIIA or IIIB NSCLC.
Time Frame: From the time of consent until 30 days after last dose of pembrolizumab up to a maximumof 18 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 92
Participants | 52

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from the time of consent until 30 days after last dose of Pembrolizumab up to a maximum of 18 months. All-Cause mortality was assessed from the date of randomization up to a maximum of 47 months or death.
Description: Adverse events were collected for every subject at every cycle of treatment (18 cycles) at an interval of 21 days from the time of consent until 30 days after last dose of Pembrolizumab.Serious adverse events and the concomitant medications used to treat them were collected up to 90 days post treatment.
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 41/93
Serious Adverse Events (participants affected / at risk) | 26/93
Other Adverse Events (participants affected / at risk) | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=93)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
AUTOIMMUNE DISORDER (Immune system disorders) | 1 (1)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
FEVER (General disorders) | 2 (2)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 7 (10)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (4)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=93)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (6)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (7)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 11 (13)
ALOPECIA (Skin and subcutaneous tissue disorders) | 7 (7)
ANEMIA (Blood and lymphatic system disorders) | 16 (24)
ANOREXIA (Metabolism and nutrition disorders) | 22 (31)
ANXIETY (Psychiatric disorders) | 20 (21)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 (29)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 (9)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (8)
ATRIAL FIBRILLATION (Cardiac disorders) | 7 (7)
AUTOIMMUNE DISORDER (Immune system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 28 (38)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 12 (18)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3)
BLURRED VISION (Eye disorders) | 4 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
BRONCHIAL INFECTION (Infections and infestations) | 5 (5)
BRONCHIAL STRICTURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 9 (9)
CATARACT (Eye disorders) | 2 (2)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
CHILLS (General disorders) | 8 (9)
CHOLESTEROL HIGH (Investigations) | 11 (12)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (2)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (2)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 27 (29)
COUGH (Respiratory, thoracic and mediastinal disorders) | 64 (124)
CREATININE INCREASED (Investigations) | 12 (25)
DEHYDRATION (Metabolism and nutrition disorders) | 8 (8)
DEPRESSION (Psychiatric disorders) | 20 (23)
DIARRHEA (Gastrointestinal disorders) | 25 (44)
DIZZINESS (Nervous system disorders) | 14 (17)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (6)
DYSGEUSIA (Nervous system disorders) | 9 (10)
DYSPEPSIA (Gastrointestinal disorders) | 6 (8)
DYSPHAGIA (Gastrointestinal disorders) | 10 (10)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 54 (97)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 5 (5)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA FACE (General disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 8 (9)
EJECTION FRACTION DECREASED (Investigations) | 2 (2)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 5 (8)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 3 (3)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 2 (2)
ESOPHAGEAL PAIN (Gastrointestinal disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 2 (2)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 6 (7)
FALL (Injury, poisoning and procedural complications) | 2 (3)
FATIGUE (General disorders) | 67 (115)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1)
FEVER (General disorders) | 14 (26)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
FLASHING LIGHTS (Eye disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
FLOATERS (Eye disorders) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 4 (5)
FLUSHING (Vascular disorders) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
GAIT DISTURBANCE (General disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 19 (20)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 9 (16)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 21 (71)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 (6)
GLAUCOMA (Eye disorders) | 2 (2)
GUM INFECTION (Infections and infestations) | 1 (1)
HEADACHE (Nervous system disorders) | 16 (19)
HEARING IMPAIRED (Ear and labyrinth disorders) | 3 (3)
HEART FAILURE (Cardiac disorders) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 8 (8)
HOT FLASHES (Vascular disorders) | 2 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 11 (14)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 37 (72)
HYPERTHYROIDISM (Endocrine disorders) | 9 (11)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 5 (7)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 11 (16)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 9 (10)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (7)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 6 (8)
HYPOTENSION (Vascular disorders) | 7 (8)
HYPOTHYROIDISM (Endocrine disorders) | 13 (19)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 2 (3)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 5 (6)
INSOMNIA (Psychiatric disorders) | 31 (34)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 4 (6)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 2 (2)
KYPHOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
LARYNGEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1)
LOCALIZED EDEMA (General disorders) | 2 (2)
LUNG INFECTION (Infections and infestations) | 5 (5)
LYMPHOCYTE COUNT DECREASED (Investigations) | 8 (18)
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 (1)
MALAISE (General disorders) | 3 (6)
MENOPAUSE (Social circumstances) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 6 (6)
MUCOSAL INFECTION (Infections and infestations) | 3 (3)
MUCOSITIS ORAL (Gastrointestinal disorders) | 4 (4)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 16 (27)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (10)
NAIL INFECTION (Infections and infestations) | 1 (1)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 12 (12)
NAUSEA (Gastrointestinal disorders) | 30 (43)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 9 (10)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 17 (23)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (4)
NON-CARDIAC CHEST PAIN (General disorders) | 9 (10)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 (2)
OTITIS EXTERNA (Infections and infestations) | 1 (2)
PAIN (General disorders) | 15 (16)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 18 (20)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 4 (4)
PELVIC PAIN (Reproductive system and breast disorders) | 2 (2)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 5 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 19 (21)
PERSONALITY CHANGE (Psychiatric disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 6 (10)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (10)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 20 (26)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 5 (6)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (21)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 17 (21)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 1 (1)
PSYCHOSIS (Psychiatric disorders) | 2 (3)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 5 (5)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 18 (35)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 8 (9)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 22 (38)
RESTLESSNESS (Psychiatric disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SINUS PAIN (Nervous system disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 6 (7)
SINUSITIS (Infections and infestations) | 6 (10)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 21 (29)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (2)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 4 (4)
SOFT TISSUE NECROSIS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 6 (6)
STROKE (Nervous system disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (4)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 4 (4)
TOOTH INFECTION (Infections and infestations) | 4 (4)
TOOTHACHE (Gastrointestinal disorders) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 6 (7)
URINARY FREQUENCY (Renal and urinary disorders) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 6 (8)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 2 (2)
URINE DISCOLORATION (Renal and urinary disorders) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 2 (2)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 2 (4)
VOMITING (Gastrointestinal disorders) | 14 (17)
WEIGHT GAIN (Investigations) | 15 (17)
WEIGHT LOSS (Investigations) | 8 (8)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 8 (10)
WHITE BLOOD CELL DECREASED (Investigations) | 7 (8)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT02343952/Prot_SAP_000.pdf